CLINICAL TRIAL: NCT04205097
Title: Deep Versus Moderate Neuromuscular Blocks on Remifentanil Requirements in Patients Undergoing Surgical Pleth Index-guided Analgesia for Laparoscopic Gastrectomy
Brief Title: Deep vs Moderate Neuromuscular Blocks on Remifentanil for Laparoscopic Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AJIRB-MED-THE-19-217
Record Dates: First submitted 2019-12-16; First posted 2019-12-19 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Neostigmine; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate NMB group (Placebo Comparator): maintaining of moderate neuromuscular block (train-of-four count 1-2) during surgery, reversal using neostigmine 50 ug/kg and glycopyrrolate 10 ug/kg
  Interventions: Drug: Neostigmine + glycopyrate
- Deep NMB group (Experimental): maintaining of deep neuromuscular block (posttetanic count 1-2) during surgery, reversal using sugammadex 2~4 mg/kg
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Neostigmine + glycopyrate — maintaining of moderate neuromuscular block (train-of-four count 1-2) during surgery, reversal using neostigmine 50 ug/kg and glycopyrrolate 10 ug/kg
  Arms: Moderate NMB group
Drug: Sugammadex — maintaining of deep neuromuscular block (posttetanic count 1-2) during surgery, reversal using sugammadex 2-4 mg/kg
  Arms: Deep NMB group

SUMMARY:
The primary purpose is to compare the remifentanil requirements in deep vs moderate neuromuscular blocks during the surgical pleth index -guided anesthesia in patients undergoing laparoscopic gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastric cancer Scheduled laparoscopic gastrectomy

Exclusion Criteria:

* Patients refusal to consent Hyperbilirubinemia Chronic pain Opioid abuse Incurrent infective status Peripheral vascular disease

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
total dose of remifentanil | from pneumoperitoneum to removal of laparoscope
  remifentanil infusion using target effect-site concentration to achieve an surgical pleth index of range between 20 and 50

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine, Suwon, Gyeonggido, South Korea